CLINICAL TRIAL: NCT07251114
Title: AI-assisted Endoscopic Ultrasound Grading of Early Esophageal Cancer Invasion Depth: A Multicenter, Prospective, Randomized Cohort Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Wei Liang, Digestive Endoscopy Center, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: K2025-02-067
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Cancer Stage; Early Esophageal Cancer
Keywords: early esophageal cancer; Artificial Intelligence; EUS
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: Use artificial intelligence to assist in the determination of the invasion depth of early esophageal squamous cell carcinoma under endoscopic ultrasound
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI Group (Experimental): Use artificial intelligence to assist in the determination of the invasion depth of early esophageal squamous cell carcinoma under endoscopic ultrasound
  Interventions: Device: Artificial Intelligence system
- Control group (No Intervention): Routine diagnosis

INTERVENTIONS:
Device: Artificial Intelligence system — Use artificial intelligence to assist in the determination of the invasion depth of early esophageal squamous cell carcinoma under endoscopic ultrasound
  Other Names: Artificial Intelligence
  Arms: AI Group

SUMMARY:
This study mainly uses an artificial intelligence system to assist in the classification of the depth of invasion of early esophageal squamous cell carcinoma under ultrasound endoscopy, providing a basis for preoperative T staging and diagnosis and treatment decisions.

DETAILED DESCRIPTION:
For patients with early esophageal squamous cell carcinoma and precancerous lesions who met the inclusion and exclusion criteria and voluntarily participated in this project, they were randomly divided into the AI group and the conventional group by central randomization, with 100 cases in each group（anticipated）. Randomization method: The personnel responsible for randomization at the center (who do not participate in the inclusion of subjects) log in to the central randomization system to obtain a randomization number, and finally form a randomization allocation table. Blinding implementation: The observation group and control group determined on the random allocation table were marked as A and B respectively, and then the operating physician implemented protocol A or B. Main indicators: Grading judgment of infiltration depth, pathological consistency

ELIGIBILITY:
Inclusion Criteria:

* Satisfy ①⑧⑨ and one of the following conditions simultaneously: ②③④⑤⑥⑦ ① Age over 18 years old, ② Esophageal ulcer, ③ low-grade intraepithelial neoplasia, ④ high-grade intraepithelial neoplasia, ⑤ patients with esophageal squamous cell carcinoma, ⑥ white patches of esophageal mucosa, ⑦ esophageal polyps, ⑧ with endoscopic examination records and detailed pathological records, ⑨ agree to participate in the study;

Exclusion Criteria:

* ① Patients who have undergone esophageal cancer surgery, ② those with a history of radiotherapy and chemotherapy for esophageal cancer, ③ patients with missing data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of grading judgment of infiltration depth | 2 years
  By comparing with the postoperative pathology, the accuracy of the preoperative T grading with the assistance of the artificial intelligence grading system was verified

SECONDARY OUTCOMES:
survival rate | Three years
  3-year survival rate
Progression Free-Survival | 1 year
  The period from the start of treatment to tumor progression or death for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Wei Liang, MD, Principal Investigator — Fujian Provincial Hospital
Locations (5):
- China (5):
  - Fujian provincial hospital, Fuzhou, Fujian
  - Affiliated Hospital of Putian University, Putian, Fujian
  - Putian First Hospital, Putian, Fujian
  - Putian Hospital of Traditional Chinese Medicine, Putian, Fujian
  - Xianyou County General Hospital, Putian, Fujian

IPD SHARING:
Plan to Share IPD: No
It involves the protection of patent technology